CLINICAL TRIAL: NCT02528591
Title: Prospective Single-center Study Evaluating the Central Blood Pressure in Renal Transplantation
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1208159; 2012-A01534-39 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Transplant
Keywords: patient; renal transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- renal transplant patient (Experimental)
  Interventions: Device: oscillometric device (Arteriograph®, Medexpert)

INTERVENTIONS:
Device: oscillometric device (Arteriograph®, Medexpert) — Central blood pressure recorded in the non-fistula arm using a validated oscillometric device (Arteriograph®, Medexpert).

SUMMARY:
The renal transplant patient is at high cardiovascular risk compared to the general population. The cardiovascular mortality represents one of the most important causes of late graft loss. Cardiovascular risk prediction tools applied to the general population, however, are caught failing on the population of kidney transplant and tend to underestimate the actual risk.

Central blood pressure is the pressure imposed at large artery (aorta, carotid) and is directly related to the target organ (heart, kidney, brain). Central blood pressure could be a cardiovascular risk factor more robust and powerful than brachial blood pressure.

Central blood pressure may in part explain the increased risk of cardiovascular disease in the population of kidney transplant patients. A cohort of 250 kidney transplant patients will be constituted with a measure of concomitant central hemodynamic monitoring to the annual review will be conducted. The main objective of this study is to describe the central blood pressure measured by oscillometric method in renal transplanted population.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Renal transplant patient

Exclusion Criteria:

* Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
central blood pressure | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARIAT, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France